CLINICAL TRIAL: NCT05296772
Title: A Phase 1 Study of JS014, a Recombinant Fusion Protein of Interleukin-21 and Humanized Anti-human Serum Albumin VHH Antibody as a Single Agent or in Combination With Pembrolizumab in Subjects With Advanced Cancer
Brief Title: Phase 1 First-in-human Study of JS014
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anwita Biosciences (Industry)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AWT-EXK21-001
Record Dates: First submitted 2022-02-28; First posted 2022-03-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Neoplasm Malignant; Neoplasm, Experimental; Solid Tumor, Adult; Lymphoma
Keywords: phase 1; JS014; first-in-human
MeSH Terms: conditions — Neoplasms; Neoplasms, Experimental; Lymphoma | interventions — Interleukin-21; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Other): A open-label single arm of JS014 alone or in combination with pembrolizumab
  Interventions: Biological: JS014, Interleukin 21 and humanized anti-human serum albumin VHH antibody; Biological: Pembrolizumab - anti-PD-1 antibody

INTERVENTIONS:
Biological: JS014, Interleukin 21 and humanized anti-human serum albumin VHH antibody — Weekly infusion at the designated dose level until disease progression, withdrawal or up to two years
Biological: Pembrolizumab - anti-PD-1 antibody — 200 mg, once every three weeks until disease progression, withdrawal or up to two years
  Other Names: Keytruda

SUMMARY:
This phase 1, first-in-human study uses a BOIN design to assess the safety and potential efficacy of JS014 at different dose levels as a single agent and in combination with fixed dose of pembrolizumab in subjects with advanced cancer.

DETAILED DESCRIPTION:
This study has two parts: 1a and Ib. Ia is a single agent study, and Ib is a combination study, testing the safety of JS014 with 200 mg of pembrolizumab. After being informed about the study and the potential risks, all subjects giving written informed consent will receive at most 4-week screening procedures to ensure the eligibility of the study entry. Once eligible, the subjects will receive JS014 infusion at the designated dose levels once every week until disease progression. In Ia study, only JS014 is given. In Ib study, JS014 will be given once a week with pembrolizumab at 200 mg once every three weeks until disease progression. The subjects will receive safety evaluation, pharmacokinetic and pharmacodynamic studies, as well as efficacy evaluation at regular interval.

The maximum number in each part of the study is 30 subjects. The Ia study will be conducted in Taiwan, and Ib study will be conducted in both Taiwan and the United States.

ELIGIBILITY:
Inclusion Criteria:

* Older 18 years of age or per local regulation
* Subjects with advanced cancer or lymphoma who have no standard therapy available, ineligible for standard therapy or unwilling to receive cytotoxic therapy .
* ECOG PS 0-1
* A life expectancy longer than three months
* Adequate organ functions
* Able to adopt effective contraceptive measures

Exclusion Criteria:

* Known history of allergies to JS014 or IL-21 or human serum albumin or pembrolizumab (Ib only)
* Subjects who have received major surgery less than 4 weeks before 1st infusion of JS014
* Subjects who has a history of immune-related adverse events in prior immunotherapy.
* Subjects who have received immunosuppressive therapy less than 4 weeks before 1st infusion of JS014.
* Subjects who have two or more primary cancers in the past 5 years.
* Newly diagnosed or symptomatic brain metastases.
* Subjects who have received prior anti-cancer therapy with residual toxicities greater than grade 2.
* Subjects who have a history of autoimmune disease in 2 years.
* Subjects who have active infection, or uncontrollable hypertension, unstable angina, active peptic ulcer, recent acute myocardial infarction, severe congestive heart failure, or unhealed wound.
* Subjects with active hepatitis B or hepatitis C.
* Subjects who are pregnant or breast feeding.
* Subjects who primary immune deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The numbers of participants with treatment-related adverse events assessed by CTCAE 5.0 | 24 months
  To determine the percentage of various toxicities assessed by CTCAE at different dose levels alone or in combination with pembrolizumab
Maximum tolerated dose (MTD) of JS014 | 24 months
  To determine the MTD of JS014 alone or in combination with pembrolizumab
Recommended phase-2 dose (RP2D) of JS014 | 24 months
  To determine of the RP2D of JS014 alone or in combination of pembrolizumab

SECONDARY OUTCOMES:
Area under the curve (AUC) of JS014 | 24 months
  To estimate the AUC of JS014 at different dose levels alone or in combination with pembrolizumab
Maximum concentration (Cmax) of JS014 | 24 months
  To measure the Cmax after 1st and repeat dose of JS014 alone or in combination with pembrolizumab
Clearance of JS014 | 24 months
  To estimate the clearance of JS014 after 1st and repeat dose of JS014 alone or in combination with pembrolizumab
Half life (T1/2) of JS014 | 24 months
  To estimate the T1/2 at terminal phase of JS014 after 1st and repeat dose of JS014 alone or in combination with pembrolizumab
Volume of distribution (Vd) of JS014 | 24 months
  To estimate Vd of JS014 after 1st and repeat dose alone or in combination with pembrolizumab
Time to reach maximum concentration (Tmax) of JS014 | 24 months
  To estimate Tmax of JS014 after 1st and repeat dose of JS014 alone or in combination with pembrolizumab
Overall response rate (ORR) alone or in combination with pembrolizumab | 24 months
  The assess the ORR of JS014 alone or in combination with pembrolizumab at different dose levels
Duration of response (DoR) alone or in combination with pembrolizumab | 24 months
  To estimate the DoR at different dose levels alone or in combination with pembrolizumab
Prevalence of anti-JS014 antibody | 24 months
  To estimate prevalence of anti-JS014 antibody at different dose levels alone or in combination with pembrolizumab
Titers of anti-JS014 antibody | 24 months
  To measure the titer of anti-JS014 antibody alone or in combination with pembrolizumab at different dose levels during the study

CONTACTS AND LOCATIONS:
Overall Officials: TJ Chiou, MD, Principal Investigator — Wanfang Hospital-Taipei Medical University
Locations (2):
- Taiwan (2):
  - Taipei Medical University -Shuang Ho Hospital, New Taipei City
  - Wanfang Hospital -Taipei Medical University, Taipei

IPD SHARING:
Plan to Share IPD: No